CLINICAL TRIAL: NCT00343980
Title: Safety and Efficacy of Inhaled Pre-prandial Human Insulin Plus Glimepiride Versus Rosiglitazone Plus Glimepiride in Type 2 Diabetes
Brief Title: Safety and Efficacy of Inhaled Pre-prandial Human Insulin in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1682
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: inhaled human insulin; Drug: glimepiride
- B (Active Comparator)
  Interventions: Drug: rosiglitazone; Drug: glimepiride

INTERVENTIONS:
Drug: rosiglitazone — Tablets, 4 mg once or twice a day.
  Arms: B
Drug: inhaled human insulin — Treat-to-target dose titration scheme, pre-prandial, inhalation.
  Other Names: NN1998
  Arms: A
Drug: glimepiride — Tablets, 4 mg/day.

SUMMARY:
This trial is conducted in Asia, Europe and Oceania. The aim of this research study is to compare the efficacy of adding inhaled preprandial insulin to glimepiride compared to adding rosiglitazone to glimepiride for the treatment of type 2 diabetes and to verify its safety (hypoglycaemia, pulmonary function, body weight, insulin antibodies and side effects)

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with OAD(s) for more than or equal to 2 months
* Body mass index (BMI) less than or equal to 40.0 kg/m2
* HbA1c greater than or equal to 8.0 % and less than or equal to 11.0 % for subjects in OAD monotherapy
* HbA1c greater than or equal to 7.5 % and less than or equal to 10.0 % for subjects on OAD combination therapy

Exclusion Criteria:

* Recurrent major hypoglycaemia
* Current smoking or smoking within the last 6 months
* Impaired hepatic or renal function
* Cardiac problems
* Uncontrolled hypertension
* Proliferative retinopathy or maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2006-10-10 (Actual); Primary Completion 2008-03-10 (Actual); Study Completion 2008-03-10 (Actual)

PRIMARY OUTCOMES:
Treatment difference in HbA1c | After 26 weeks

SECONDARY OUTCOMES:
Adverse events | For the duration of the trial
Body weight | during treatment
Lung function | after 26 weeks of treatment
Blood glucose | after 26 weeks of treatment
Hypoglycaemia | from 12-26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (20):
- Australia (4):
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Garran
  - Novo Nordisk Investigational Site, Kingswood
- Croatia (2):
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Zagreb
- India (5):
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Bangalore
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Coimbatore
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Philippines (3):
  - Novo Nordisk Investigational Site, Cebu City
  - Novo Nordisk Investigational Site, Makati City
  - Novo Nordisk Investigational Site, Manila
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Bursa
  - Novo Nordisk Investigational Site, Istanbul

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com